CLINICAL TRIAL: NCT03809585
Title: Observational Study of Iris Tumors
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, Peterson Professor of Ophthalmology & Professor of Biomedical Engineering, Oregon Health and Science University
Other Study IDs: 6612-IRIS; R01EY028755 (NIH)
Record Dates: First submitted 2018-11-29; First posted 2019-01-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Iris Tumor
Keywords: Iris; Tumor; Melanoma; Optical Coherence Tomography (OCT); Angiography
MeSH Terms: conditions — Iris Neoplasms; Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Iris Tumors: This group will consist of 50 adults age 18 or older who have been diagnosed with either melanotic or amelanotic iris tumors. Iris tumor diagnosis will be confirmed by biopsy when possible or based upon clinical features (if patient declines biopsy or if not medically indicated) according to standard-of-care guidelines.
- Healthy Controls: This group will consist of 50 adults age 18 and older who have healthy eyes.

SUMMARY:
This is an observational study using OCT angiography to assist with tumor characterization in melanotic and amelanotic iris lesions. OCT angiography data from healthy eyes will be compared to eyes with various types of iris tumors.

ELIGIBILITY:
Inclusion Criteria for tumor group:

* Eyes with diagnosis of melanotic or amelanotic iris tumors

Inclusion Criteria for healthy control group:

* Eyes without iris defects or lesions

Exclusion Criteria (both groups):

* Inability to give informed consent
* Inability to maintain stable fixation for OCT imaging
* Inability to commit to required study visits
* Eyes with concurrent retinal diseases, glaucoma, or conditions that in the opinion of the investigators might affect iris circulation
* Mature cataracts if found to limit visual potential to worse than 20/40

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults age 18 or older with either healthy eyes or iris tumors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Tumor Thickness in Benign vs Malignant Iris Lesions | 6 months
  OCT/OCTA will be used to compare tumor thickness measurements against the conventional Ultrasonic Biomicroscopy (UBM) device. Tumor thickness will be measured in millimeters, and growth of 0.5 mm or greater will be used to differentiate malignant from benign lesions.

SECONDARY OUTCOMES:
Tumor Area in Benign vs Malignant Iris Lesions | 6 months
  Tumor area will be measured by OCT/OCTA in mm2 and compared against conventional UBM measurements.
Tumor Volume in Benign vs Malignant Iris Lesions | 6 months
  Tumor volume will be measured by OCT/OCTA in mm3 and compared against conventional UBM measurements.
Effect of Radiation Treatment on Tumor and Surrounding Ocular Structures | 6 months after treatment
  Vessel density and tortuosity will both be measured in % occupied by flow pixels on OCT/OCTA.

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States